CLINICAL TRIAL: NCT02456649
Title: A Phase II Study of the Outcomes of Intraoperative Margin Assessment With Adjunctive Use of MarginProbe in Addition to Standard
Brief Title: Study of the Outcomes of Intraoperative Margin Assessment With MarginProbe
Acronym: MarginProbe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huntington Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jeannie Shen, Medical director, Breast Surgery, Huntington Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HMH2015.001
Record Dates: First submitted 2015-05-19; First posted 2015-05-28 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer
Keywords: lumpectomy margins
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MarginProbe (Experimental): Single arm study - MarginProbe in addition to standard procedure
  Interventions: Device: MarginProbe

INTERVENTIONS:
Device: MarginProbe — Intraoperative MarginProbe use as adjunct to standard practice MarginProbe will be used on the lumpectomy specimen within 20 minutes of excision, prior to specimen Xray or gross pathology evaluation. This may take up to 5 minutes. MarginProbe will indicate a positive or negative reading for each of the 6 circumferential margins, and the results will be recorded. Any margins determined by to < 5-10 mm by specimen Xray or gross pathology examination will be re-excised. In addition, any additional margins not already identified as < 5-10 mm, but identified as positive by MarginProbe will be re-excised where feasible.

SUMMARY:
The combination of breast conserving surgery (lumpectomy) with radiation therapy has been shown to result in equivalent overall survival rates compared to mastectomy for the local treatment of breast cancer. As a result, the majority of patients diagnosed with breast cancer in the United States undergo lumpectomy as their primary surgical therapy. Multiple studies have demonstrated the association between positive lumpectomy margins and an increased risk of ipsilateral breast tumor recurrence, even with postoperative radiation. Studies report 20-40% of lumpectomy procedures result in one or more involved (positive) surgical margins, leading to the need for further surgery, emotional distress, poorer cosmesis, delay to adjuvant treatments, and increased cost. Current available intraoperative margin assessment techniques include specimen Xray, gross pathology, frozen section, and touch prep cytology. To reduce the incidence of positive margins, the MarginProbe (Dune Medical Devices, Caesarea, Israel) was developed to provide real-time, intraoperative assessment of the presence of tumor at the lumpectomy margin. In the current study, the investigators aim to determine the effectiveness of MarginProbe as an adjunctive tool to standard practice for intraoperative identification of tumor at lumpectomy margins, and its ability to reduce positive margins and decrease the need for additional surgical procedures.

DETAILED DESCRIPTION:
In the current study, the investigators aim to determine the effectiveness of MarginProbe as an adjunctive tool to standard practice for intraoperative identification of tumor at lumpectomy margins, and its ability to reduce positive margins and decrease the need for additional surgical procedures.

Aims of the study:

Primary objectives

1. Determine positive margin rate following lumpectomy

Secondary objectives

1. Determine accuracy of intraoperative margin assessment with use of MarginProbe plus standard of care (gross pathologic examination and/or intraoperative specimen Xray) versus standard of care (gross pathologic examination and/or intraoperative specimen Xray) alone.
2. Determine impact of MarginProbe on total tissue volume removed
3. Determine the impact of MarginProbe on the need for additional surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects able to read and understand the informed consent

Exclusion Criteria:

1. Subjects unable to read or understand the informed consent.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with histologically positive surgical margins | 2 weeks after surgery

SECONDARY OUTCOMES:
Percentage of patients who undergo a second surgery after initial lumpectomy. | 2 weeks after surgery
False positive and false negative rate of Intraop MarginProbe results compared to histologic evaluation | 2 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jeannie Shen, MD, Principal Investigator — Huntington Memorial Hospital
Locations (1):
- Huntington Memorial Hospital, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moran MS, Schnitt SJ, Giuliano AE, et al. JCO Feb 10, 2014.
- [Result] Allweis TM, Kaufman Z, Lelcuk S, Pappo I, Karni T, Schneebaum S, Spector R, Schindel A, Hershko D, Zilberman M, Sayfan J, Berlin Y, Hadary A, Olsha O, Paran H, Gutman M, Carmon M. A prospective, randomized, controlled, multicenter study of a real-time, intraoperative probe for positive margin detection in breast-conserving surgery. Am J Surg. 2008 Oct;196(4):483-9. doi: 10.1016/j.amjsurg.2008.06.024. PMID 18809049
- [Result] Pappo I, Spector R, Schindel A, Morgenstern S, Sandbank J, Leider LT, Schneebaum S, Lelcuk S, Karni T. Diagnostic performance of a novel device for real-time margin assessment in lumpectomy specimens. J Surg Res. 2010 May 15;160(2):277-81. doi: 10.1016/j.jss.2009.02.025. Epub 2009 Mar 31. PMID 19628225
- [Result] Rivera RJ, Holmes DR, Tafra L. Analysis of the Impact of Intraoperative Margin Assessment with Adjunctive Use of MarginProbe versus Standard of Care on Tissue Volume Removed. Int J Surg Oncol. 2012;2012:868623. doi: 10.1155/2012/868623. Epub 2012 Dec 26. PMID 23326653
- [Result] Thill M, Dittmer C, Baumann K, Friedrichs K, Blohmer JU. MarginProbe(R)--final results of the German post-market study in breast conserving surgery of ductal carcinoma in situ. Breast. 2014 Feb;23(1):94-6. doi: 10.1016/j.breast.2013.11.002. Epub 2013 Dec 2. PMID 24291375
- [Result] Schnabel F, Boolbol SK, Gittleman M, Karni T, Tafra L, Feldman S, Police A, Friedman NB, Karlan S, Holmes D, Willey SC, Carmon M, Fernandez K, Akbari S, Harness J, Guerra L, Frazier T, Lane K, Simmons RM, Estabrook A, Allweis T. A randomized prospective study of lumpectomy margin assessment with use of MarginProbe in patients with nonpalpable breast malignancies. Ann Surg Oncol. 2014 May;21(5):1589-95. doi: 10.1245/s10434-014-3602-0. Epub 2014 Mar 5. PMID 24595800
- [Result] Police AM. Routine use of a real time margin assessment device. Poster Abstract presented at the 31st Annual Miami Breast Cancer Conference; May 2014.
- [Result] Sebastian M, Akbari S. Combined experience at three breast centers with routine use of an intraoperative margin assessment device including comparison to historical re-excision rates. Poster Abstract presented at ASCO Breast Cancer Symposium; September 2014.